CLINICAL TRIAL: NCT03396887
Title: The Effectiveness of a Smartphone Application in the Treatment of Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Patrick's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr. Conor Farren, Consultant Psychiatrist, St Patrick's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCD - Protocol 19/15
Record Dates: First submitted 2017-05-12; First posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-11

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Smartphone Application
MeSH Terms: conditions — Alcoholism | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to intervention or control condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application Users (Experimental): The experimental group will receive the smartphone intervention along with treatment as usual for 3-months. The smartphone application (UControlDrink) includes twice daily text message recovery support, relapse prevention cognitive behavioural therapy, 12 sessions in total, drinking and recovery activity logs where participants detail their abstinence, drinking and recovery activity engagement on a daily basis. Craving intervention in the form of a "calm button" to deal with cravings and prevent relapse and gamification, a system of encouraging positive behaviour with the awarding of "points" to achieve various "status" levels, is used to increase adherence and compliance with treatment recommendations.
  Interventions: Other: U Control Drink Smartphone Application
- Control Group (Active Comparator): The control group will also receive treatment as usual, i.e. any follow-up after-care that they chose to participate in and regular AA/Lifering meetings.
  Interventions: Other: Control group

INTERVENTIONS:
Other: U Control Drink Smartphone Application — The smartphone application comprises five recovery focused features: supportive messages, Computerised-Cognitive Behavioural Therapy, a drinking log, craving management and gamification.
  Arms: Smartphone Application Users
Other: Control group — The control group will receive treatment as usual.
  Arms: Control Group

SUMMARY:
Alcohol dependence poses a major problem for Irish and UK society, placing a huge burden on the health system. It is difficult to treat and relapse is common. There is an urgent need to develop novel treatment methods. One growing area of intervention is the use of mobile phone technology to develop personalised, patient-centred treatments. These can be used in outpatient settings, allowing patients to manage their own illness and take control of their recovery. In this study the investigators will investigate how a smartphone application, UControlDrink, can help alcoholics stay abstinent from alcohol. The application consists of a number of features known to aid recovery such as supportive messages and online therapy.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a common and difficult disorder to treat. Only a fraction of sufferers seek treatment and the rate of relapse is high. There is therefore an urgent need for improved methods of promoting long term abstinence and recovery in AUD. This study will explore the effectiveness of a smartphone application, UControlDrink, in aiding recovery from AUD in patients who have been discharged from an inpatient alcohol treatment programme. The application comprises five recovery focused features:

supportive messages, Computerised-Cognitive Behavioural Therapy, a drinking log, activities and trigger avoidance log, craving management and gamification. Patients will use the application for 3 months. A control group of patients will also be followed over the same time period. Cumulative abstinence duration as well as changes in questionnaire measures to baseline, time to first drink, proportion of patients continuously abstinent from alcohol, levels of activity within the app and patient satisfaction with their overall treatment will be measured at 3 months. If successful, this application may offer a unique, patient-centred, technology-driven, cost effective method of improving outcomes in AUD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will fulfil the criteria for an alcohol use disorder according to the Structured Clinical Interview for DSM-5 Axis I Disorders
2. Patients must complete an alcohol treatment programme at St. Patrick's University Hospital.
3. Primary addiction must be alcohol in poly-substance abusers.
4. Aged over 18 years of age and capable of providing written, informed consent.
5. Mini Mental State Examination (MSSE) score of ≥25.
6. Patients must have an iphone or Android smartphone and are familiar with using smartphone applications.

Exclusion Criteria:

1. Patients whose primary substance of abuse is not alcohol, although may meet the criteria for alcohol dependency/abuse.
2. Patients who do not have an iPhone or Android smartphone.
3. Age <18years or >70years.
4. Psychotic disorder
5. Patients who do not fully complete an inpatient treatment programme before discharge.
6. History of alcohol use disorder but not current.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of drinking days | 3 months
  The number of drinking days will be assessed using the Time Line to Follow-Back scale (TLFB).The Alcohol TLFB is a descriptive questionnaire, using a calendar, participants will retrospectively record the number of days they drank over the previous 90 days. Drinking days will be calculated by summing the total number of days when alcohol was consumed in the previous 90 days.
App activity score | 3 months
  Activity score on the app
Units of alcohol consumed per drinking day | 3 months
  The Time Line Follow Back (TLFB) will be used to record the average number of units of alcohol consumed on drinking days.

SECONDARY OUTCOMES:
Time to first drink | 3 months
  Number of days to first drink
Changes in the Alcohol Use Disorders Identification Test scores from baseline | 3 months
  Changes in scores on the Alcohol Use Disorders Identification Test between baseline and 3 month follow-up assessment.
Changes in the Alcohol Abstinence Self-Efficacy Scale scores from baseline | 3 months
  Changes in the Alcohol Abstinence Self-Efficacy Scale scores between baseline and 3 month follow-up assessment.
Changes in the Obsessive Compulsive Drinking Scale scores from baseline | 3 months
  Changes in scores on the Obsessive Compulsive Drinking Scale between baseline and 3 month follow-up assessment.
Changes in the Beck Depression Inventory scores from baseline | 3 months
  Changes in scores on the Beck Depression Inventory between baseline and 3 month follow-up assessment.
Changes in the Beck Anxiety Inventory scores from baseline | 3 months
  Changes in scores on the Beck Anxiety Inventory between baseline and 3 month follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Farren, PhD,MRCPsych, Principal Investigator — St. Patrick's University Hospital
Locations (1):
- St. Patrick's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No